CLINICAL TRIAL: NCT07286500
Title: "Impact of Sexual Activity on Hypoglycemia Risk in Adults With Type 1 and Type 2 Diabetes Under Insulin Therapy and Continuous Glucose Monitoring (CGM)"
Brief Title: "Sexual Activity and Hypoglycemia Risk in Adults With Type 1 or Type 2 Diabetes Using Insulin Therapy and Continuous Glucose Monitoring"
Acronym: SEX-HYPO-CGM
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Collaborators: Jagiellonian University Medical College - Department and Clinic of Metabolic Diseases (Katedra i Klinika Chorób Metabolicznych UJ) (Unknown)
Responsible Party: Sponsor
Other Study IDs: KB/112/2025
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes (T1D); Type 2 Diabetes (T2DM); Hypoglycemia
Keywords: Sexual Activity; Hypoglycemia; Glucose Variability; Continuous Glucose Monitoring; CGM; Insulin Therapy; Type 1 Diabetes; Type 2 Diabetes; Diabetes Complications
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Hypoglycemia; Sexual Behavior; Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetes Cohort: Adults with type 1 or type 2 diabetes treated with insulin therapy and using continuous glucose monitoring (CGM). Participants are observed for 3 months. They mark sexual activity in their CGM application, and glucose values during and up to 6 hours after the activity are analyzed and compared with glucose data from days without sexual activity.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study. No intervention is assigned. Participants continue their usual insulin therapy and self-management. Sexual activity is self-initiated and only marked within the CGM application for observational purposes

SUMMARY:
This observational study examines whether sexual activity influences the risk of hypoglycemia in adults with type 1 or type 2 diabetes treated with insulin therapy and using continuous glucose monitoring (CGM). Many patients report fear of hypoglycemia during or after sexual activity, which may affect their quality of life and willingness to engage in intimate relationships. However, no systematic research has been conducted on this topic, largely due to the sensitive nature of sexual health and the previous lack of tools to remotely monitor glucose profiles.

The study uses CGM systems (LibreView or Dexcom Clarity) to evaluate glucose changes during and up to 6 hours after sexual activity. Participants will mark the start of sexual activity in their CGM application using a neutral symbol (such as a heart icon). Data will be collected remotely through secure, certified platforms without the need for discussing details of intimate life. Glucose profiles from days with and without sexual activity will be compared. Each participant will be observed for 3 months.

The study will include 100 adults with type 1 or type 2 diabetes who use CGM and insulin therapy. By analyzing episodes of glucose levels below 70 mg/dL during or after sexual activity, the study aims to determine whether sexual activity is associated with an increased risk of hypoglycemia. Findings may help to better understand patient concerns, reduce unnecessary fear, and develop future clinical recommendations for safe sexual activity in individuals treated with insulin.

DETAILED DESCRIPTION:
Sexual health is an integral component of overall well-being and quality of life, including for adults living with chronic diseases such as diabetes. Despite its importance, sexual health is often overlooked in clinical practice. Health care professionals rarely initiate conversations about sexual functioning due to limited training, lack of tools, or concern about patient discomfort. At the same time, many patients with diabetes report fear of hypoglycemia during or after sexual activity, and partners frequently share similar concerns. These fears may lead to reduced sexual activity and diminished quality of life.

Hypoglycemia remains one of the most common and clinically significant complications of insulin therapy. Glucose levels below 70 mg/dL require prompt intake of carbohydrates or adjustment of glucose-lowering treatment to prevent further decline. Physical exertion- including sexual activity-may lead to early or delayed hypoglycemia, occurring even several hours after the activity. On the other hand, emotional excitement during sexual activity may trigger counter-regulatory hormones such as adrenaline or cortisol, potentially causing hyperglycemia. Despite these observations, no systematic study has evaluated the relationship between sexual activity and glucose fluctuations in adults with diabetes. Historically, such research was hindered by the intimate nature of the subject and the absence of remote monitoring tools.

The introduction of continuous glucose monitoring (CGM) systems, together with cloud-based platforms such as LibreView and Dexcom Clarity, enables the remote and secure assessment of glucose trends without requiring direct discussion of intimate details. This study leverages these technologies to evaluate whether sexual activity increases the risk of hypoglycemia in adults with type 1 or type 2 diabetes treated with insulin.

Each participant will be observed for 3 months. Participants will mark the beginning of sexual activity within their CGM application using a neutral icon (e.g., a heart symbol). Glucose trends during and for up to 6 hours following the activity will be analyzed and compared to glucose profiles from days without sexual activity. Health care providers will also complete a brief online form with basic clinical information about each participant, including age, diabetes type, disease duration, treatment regimen, and CGM system used.

The study aims to enroll 100 adults. This pragmatic sample size reflects the exploratory nature of the project and the absence of prior research in this area. Based on general population estimates, participants are expected to report an average of approximately 10 episodes of sexual activity over the 3-month observation period. The primary endpoint is the proportion of sexual activity episodes associated with hypoglycemia, defined as glucose levels below 70 mg/dL occurring during or after the activity.

All data will be anonymized. Each patient will receive a unique study code that does not contain personal identifiers. Only the principal investigator and scientific supervisor will have access to the code key. Glucose data and sexual activity markers will be exported from CGM applications in encrypted form and analyzed exclusively in de-identified datasets. After completion of the study and statistical analysis, all data will be securely deleted according to institutional procedures.

The results of this study may provide the first empirical evidence on the relationship between sexual activity and hypoglycemia risk in individuals using insulin therapy. If a relationship is confirmed, the findings may guide future recommendations to improve safety around sexual activity. If no association is found, the results may help reduce unnecessary anxiety among patients and improve open communication in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.
* Diagnosis of type 1 or type 2 diabetes.
* Current use of a continuous glucose monitoring (CGM) system.
* Treatment with insulin therapy in any regimen.
* Ability to operate the CGM application and mark the start of sexual activity.
* Willingness to participate for 3 months.
* Signed informed consent.

Exclusion Criteria:

* Inability to independently use the CGM application.
* No sexual activity during the study period.
* Withdrawal of consent at any time.
* Any condition that, in the opinion of the investigator, prevents safe participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with type 1 or type 2 diabetes who use continuous glucose monitoring (CGM) and insulin therapy. Participants will be recruited from diabetes clinics and outpatient practices. All participants must be willing to record sexual activity in the CGM application and share anonymized CGM data for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of Sexual Activity Episodes Associated With Hypoglycemia | 3 months per participant
  Hypoglycemia is defined as a glucose value below 70 mg/dL occurring during sexual activity or within 6 hours after its completion. Episodes will be identified through CGM data, using participant-marked sexual activity timestamps. Each sexual activity event will be analyzed for the presence or absence of hypoglycemia, and the proportion of events associated with hypoglycemia will be calculated.

SECONDARY OUTCOMES:
Frequency of Hypoglycemia on Sexual Activity Days vs. Non-Activity Days | 3 months per participant
  Comparison of the number of hypoglycemic episodes (glucose <70 mg/dL) during sexual activity and within 6 hours afterward versus matched time intervals on days without sexual activity. Glucose values will be obtained from CGM reports.
Mean Glucose Level During and After Sexual Activity | 3 months per participant
  Mean interstitial glucose during sexual activity and up to 6 hours after its completion, compared with mean glucose levels on matched control days without sexual activity, based on CGM data.

OTHER OUTCOMES:
Number of Sexual Activity Episodes Recorded per Participant | 3 months per participant
  Total number of sexual activity episodes marked by each participant in the CGM application during the 3-month observation period. This serves as a feasibility and compliance indicator for event recording in a sensitive clinical context.
Proportion of Participants Completing the Full Observation Period With at Least One Recorded Sexual Activity Episode | 3 months per participant
  Proportion of enrolled participants who complete the 3-month observation period and record at least one episode of sexual activity in the CGM app. This outcome assesses feasibility, retention, and participant engagement.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, CSK UCK, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamiński M, et al. Glycemic variability and clinical outcomes in diabetes. Int J Angiol. 2022;31(2):97-106. PMID: 35173854.
- [Background] Weinberg AE, Eisenberg M, Patel CJ, Chertow GM, Leppert JT. Diabetes severity, metabolic syndrome, and the risk of erectile dysfunction. J Sex Med. 2013 Dec;10(12):3102-9. doi: 10.1111/jsm.12318. Epub 2013 Sep 9. PMID 24010555
- [Background] Bąk E, et al. Sexual functioning in men and women with diabetes. Int J Environ Res Public Health. 2017;14(9):1073. PMID: 28926963.
- [Background] Cichocka E, Jagusiewicz M, Gumprecht J. Sexual Dysfunction in Young Women with Type 1 Diabetes. Int J Environ Res Public Health. 2020 Jun 22;17(12):4468. doi: 10.3390/ijerph17124468. PMID 32580278
- [Background] Buskoven MEH, Kjorholt EKH, Strandberg RB, Softeland E, Haugstvedt A. Sexual dysfunction in women with type 1 diabetes in Norway: A qualitative study of women's experiences. Diabet Med. 2022 Jul;39(7):e14856. doi: 10.1111/dme.14856. Epub 2022 Apr 28. PMID 35460298
- [Background] Winkley K, Stahl D, Kar P. Diabetes distress in adults with type 1 diabetes: A systematic review and meta-analysis. Diabet Med. 2021;38(11):e14644. PMID: 34143273.